CLINICAL TRIAL: NCT05135676
Title: Time in Glucose Hospital Target (TIGHT) - A Randomized Clinical Trial to Evaluate the Use of CGM to Achieve a Mean Glucose Target of 90 to 130 mg/dL Without Hypoglycemia in Hospitalized Adults With Type 2 Diabetes
Brief Title: Time in Glucose Hospital Target
Acronym: TIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIGHT
Record Dates: First submitted 2021-10-21; First posted 2021-11-26 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Continuous glucose monitoring; Hypoglycemia; Glycemia; Hyperglycemia; In-patient; Hospital
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Target Group (Active Comparator): Standard therapy with glucose target 140-180 mg/dL (ADA guidelines) and masked CGM
  Interventions: Device: Blinded CGM
- Intensive Target Group (Experimental): Intensive therapy with glucose target 90-130 mg/dL with real-time CGM
  Interventions: Device: real-time CGM

INTERVENTIONS:
Device: Blinded CGM — A masked CGM sensor will be worn
  Other Names: Commercially available Dexcom CGM
  Arms: Standard Target Group
Device: real-time CGM — An unmasked CGM sensor will worn
  Other Names: Commercially available Dexcom CGM
  Arms: Intensive Target Group

SUMMARY:
Inpatient management of glycemia in people with diabetes has been inadequately studied. Previous randomized trials of intensive insulin therapy in the hospital setting resulted in excessive hypoglycemia. Current ADA guidelines (glucose 140-180 mg/dL) are by consensus with the upper bound defined by observational data and the lower bound by safety concerns. None of the previous studies of intensive glucose management used CGM technology. Whether near normal glucose levels can be achieved without increasing hypoglycemia among hospitalized patients with diabetes with the advent of CGM technology is not known.

There are clear associations between hyperglycemia and poor outcomes in patients with diabetes hospitalized with infection, including COVID-19. The COVID-19 pandemic has increased the urgency to definitively answer the question of whether glucose lowering below 140-180 mg/dL can be achieved without increasing hypoglycemia.

If this proposed study demonstrates intensive management of glucose to a target of 90 to 130 mg/dL without hypoglycemia is achievable in the inpatient setting with CGM technology, a larger study could then be performed to evaluate whether there is clinical benefit including a reduction in morbidity and mortality.

The primary study hypothesis is that glucose management with CGM can achieve a mean glucose of 90-130 mg/dL without increasing hypoglycemia compared with standard care with a glucose target of 140-180 mg/dL. Individuals with diabetes who are hospitalized (non-ICU) for an eligible condition will be randomly assigned to receive standard therapy (glucose target 140-180 mg/dL per ADA guidelines) or intensive therapy (glucose target 90-130 mg/dL and CGM used for monitoring). Real-time CGM will be used in the Intensive Target Group and masked CGM will be used in the Standard Target Group.

The co-primary outcomes, assessed via a hierarchical approach, include a treatment group comparison of mean glucose (superiority) followed by a non-inferiority comparison of time <54 mg/dL measured with CGM.

DETAILED DESCRIPTION:
Protocol Overview:

* The glucose management team (GMT) at each site will identify potentially eligible patients.
* After informed consent and confirmation of eligibility, each participant will be randomly assigned to the Standard Target or Intensive Target group.
* Glucose management in the Standard Target Group will follow the hospital's usual practice using insulin for glucose management, with a target glucose concentration of 140-180 mg/dL.

  - A masked CGM sensor will be worn.
* Glucose management in the Intensive Target Group will include close monitoring by the site GMT to maximize the percentage of glucose values in the range of 90 to 130 mg/dL.

  * Glucose monitoring will include real-time CGM. The hospital's GMT will be the ones monitoring the CGM data. The information from CGM will be used for future management changes to insulin delivery and for safety monitoring, particularly for hypoglycemia. In essence, CGM will be used adjunctively in the study.
  * CGM validation will occur within 2-6 hours following sensor insertion and must be within 20% of a blood glucose result of >100 mg/dL for two consecutive blood glucose measurements. If a blood glucose result is <100 mg/dL, the corresponding CGM reading must be within 20 mg/dL of the blood glucose value. CGM validation will occur at least twice daily.
* Insulin delivery will be based on the site's usual protocol. The hospital nursing staff will follow their institutional SOPs with respect to frequency of BGM testing and use of BG test results for administering meal insulin and corrections. The nursing staff will not be utilizing CGM in this regard.
* Study participation will conclude at the time of hospital discharge, 10 days after randomization, at time of transfer to ICU or death.

Quality Assurance Plan:

Designated personnel from the Coordinating Center will be responsible for maintaining quality assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is conducted and data are generated, documented and reported in compliance with the protocol, Good Clinical Practice (GCP) and the applicable regulatory requirements, as well as to ensure that the rights and wellbeing of trial participants are protected and that the reported trial data are accurate, complete, and verifiable. Eligibility, informed consent, data entry completion and adverse events will be prioritized for monitoring.

Source Data Verification:

Study data will be obtained from the participant, the participant's EHR and from CGM. EHR data will be either transcribed from the EHR onto eCRFs on the study website or will be electronically transmitted to the Coordinating Center.

Standard Operating Procedures:

1. Patient Recruitment and Enrollment:

   Recruitment will involve identification of hospitalized patients at each clinical center who meet the study eligibility criteria. There will be no specific efforts to promote recruitment other than making hospital staff aware of the study.

   Enrollment will proceed with the goal of at least 120 participants entering the randomized trial but no greater than 150. Screening for eligibility will be performed from medical records prior to informed consent being signed. Thus, once informed consent is signed, randomization will proceed quickly. Participants who have signed consent may be permitted to continue into the trial, if eligible, even if the randomization goal has been reached.

   Study participants will be recruited from 3-6 clinical centers in the United States. All eligible participants will be included without regard to sex, race, or ethnicity. There is no restriction on the number of participants to be enrolled by each site toward the overall recruitment goal.
2. Data Collection and Testing:

   * After informed consent has been signed, all potential participants who are females of child-bearing potential will have a serum or urine pregnancy test if one has not been done since hospital admission.
   * Data from the EHR will be recorded in the study database. Medical history information will include diabetes history, other medical conditions, medications, height and weight, HbA1c (during hospitalization or most recent prior to admission), and other relevant laboratory values. The medical condition that prompted hospital admission will be recorded.
3. Data Recorded for Study (in addition to data collected at enrollment):

   At the end of hospitalization or 10 days from randomization, data to be recorded will include:
   * Vitals (blood pressure, heart rate, temperature, and O2 saturation if oxygen is used)
   * BGM
   * Insulin received each day: type of insulin, route (IV or SQ), # of units
   * All medical conditions that developed during the hospitalization
   * Date of transfer to ICU
   * Medications received
   * All coded discharge diagnoses including alive or dead
   * Labs (if measured/available) such as:

     * At admission and prior to randomization (if available)

       * Hematocrit and hemoglobin
       * Electrolytes (sodium, potassium, bicarbonate)
       * Liver function (ALT)
       * COVID-19 testing
     * All measurements (at admission and while active in the study)

       * Glucose
       * HbA1c
       * Creatinine/eGFR
4. Reporting for Adverse Events:

SAEs possibly related to a study device or study participation and UADEs must be reported to the Coordinating Center within 24 hours of the site becoming aware of the event. This can occur via phone or email, or by completion of the online serious adverse event form and device issue form if applicable. If the form is not initially completed, it should be competed as soon as possible after there is sufficient information to evaluate the event. All other reportable ADEs and other reportable AEs should be submitted by completion on the on line form within 7 days of the site becoming aware of the event. The Coordinating Center will notify all participating investigators of any adverse event that is serious, related, and unexpected. Notification will be made within 10 working days after the Coordinating Center becomes aware of the event. Each principal investigator is responsible for reporting serious study-related adverse events and abiding by any other reporting requirements specific to his/her Institutional Review Board or Ethics Committee. Where the JCHR IRB is the overseeing IRB, sites must report all serious, related adverse events within seven calendar days. Upon receipt of a qualifying event, the Sponsor will investigate the event to determine if a UADE is confirmed, and if indicated, report the results of the investigation to all overseeing IRBs, and the FDA within 10 working days of the Sponsor becoming aware of the UADE per 21CFR 812.46(b). The Medical Monitor must determine if the UADE presents an unreasonable risk to participants. If so, the Medical Monitor must ensure that all investigations, or parts of investigations presenting that risk, are terminated as soon as possible but no later than 5 working days after the Medical Monitor makes this determination and no later than 15 working days after first receipt notice of the UADE.

Sample Size:

Sample size has been computed for the treatment group comparison of mean glucose:

A total sample size was computed to be N=110 for the following assumptions: two randomized arms, 90% power, a 25 mg/dL difference in mean glucose between treatment groups, SD of 40 mg/dL, and 2-sided type 1 error of 0.05.

The total sample size has been increased to N=150 to account for potential dropouts and incomplete CGM glucose data due to early hospital discharge.

For percent of time < 54 mg/dL, statistical power will be >99% for demonstrating non-inferiority: two randomized arms, a total sample size of N=110, a standard deviation of 1%, no difference, and alpha =0.025.

Statistical Analysis Plan:

The trial has co-primary outcomes measured using CGM for up to 10 days following randomization; mean glucose tested between groups for superiority and % time <54 mg/dL tested to demonstrate non-inferiority of intensive treatment compared with standard treatment. The intervention will be considered effective only if both endpoints are met.

The null/alternative hypotheses are:

1. Mean Glucose

   1. Null Hypothesis: There is no difference in mean glucose between Standard and Intensive groups.
   2. Alternative Hypothesis: The mean glucose is different in the Standard and Intensive groups.
2. Percent Time <54 mg/dL

   1. Null Hypothesis: There is an absolute mean difference of at least 1% in the percent time <54 mg/dL between the Intensive and Standard group.
   2. Alternative Hypothesis: There is an absolute mean difference of less than 1% in the percent time <54 mg/dL between the Intensive and Standard groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years old
2. Type 2 diabetes (per investigator assessment); or if not previously diagnosed as having diabetes, HbA1c>=7.0% (laboratory-measured at or since hospital admission or within prior 3-months).

   • Type 1 diabetes, atypical forms of diabetes (including pancreatectomy and pancreatitis) and stress hyperglycemia alone are not eligible.
3. At least 1 blood glucose measurement >180 mg/dL since admission
4. Insulin already initiated since admission or planned to be initiated
5. Non-critical hospitalization with expected length of stay on non-ICU floor >3 days at time of randomization

Exclusion Criteria:

1. Inability to provide written consent
2. Admission to ICU

   • Patients transferred from ICU with an expected length of stay >3 days on a non-ICU floor are eligible
3. Treatment with systemic immunosuppressive agents such as high dose (>7.5 mg/day Prednisone equivalent) steroids or biologics that are not regimented and have been started within the last 3 months at time of enrollment or planned treatment prior to randomization.
4. Suspected or confirmed acute myocardial infarction or stroke as reason for hospital admission or since admission
5. Considered unlikely to survive hospitalization per investigator's judgment
6. Diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic state (HHS) in the 6 months prior to hospital admission, at hospital admission or prior to randomization during the current hospital admission
7. One or more severe hypoglycemic events within the 6 months prior to hospital admission or prior to randomization during the current admission
8. For females, pregnant or breastfeeding

   • A negative serum or urine pregnancy test will be required for all females of child-bearing potential.
9. CGM other than study CGM being used during hospitalization or planned to be used
10. Blood glucose >400 mg/dL at time of potential enrollment (most recent blood glucose measurement in hospital)
11. Insulin pump being used to deliver insulin during hospitalization or planned to be used
12. Use of IV insulin at time of potential enrollment
13. Hypoxia (O2 saturation <90) present at time of potential enrollment
14. Anasarca present at time of potential enrollment
15. Use of hydroxyurea or high dose acetaminophen use of >4g daily
16. eGFR <20 mL/min or dialysis being received or planned
17. ALT >3X normal or current diagnosis of cirrhosis
18. Cystic fibrosis
19. Expected need for surgery requiring general anesthesia during hospitalization

    • Post-surgical enrollment is permitted
20. Known allergy to medical grade adhesives or a skin condition that may impact CGM performance per investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Co-primary Outcome: CGM-measured mean glucose (superiority) | 4-10 days
  In this trial, one of the co-primary outcomes measured using CGM for up to 10 days following randomization is the mean glucose which is tested for superiority between the intensive treatment and standard treatment.
Co-primary Outcome: CGM-measured percent time <54 mg/dL (non-inferiority) | 4-10 days
  In this trial, the other co-primary outcome measured using CGM for up to 10 days following randomization is the percent time below 54 mg/dL which is tested to demonstrate non-inferiority of intensive treatment compared with standard treatment.

SECONDARY OUTCOMES:
CGM Metrics by daytime only (06:00 AM to 00:00 AM) | 4-10 days
  * Percent time in range 70-180 mg/dL
  * Percent time in range 70-140 mg/dL
  * Percent time above 180 mg/dL
  * Percent time above 250 mg/dL
  * Percent time below 54 mg/dL (superiority)
CGM Metrics by nighttime only (00:00 AM to 06:00 AM) | 4-10 days
  * Percent time in range 70-180 mg/dL
  * Percent time in range 70-140 mg/dL
  * Percent time above 180 mg/dL
  * Percent time above 250 mg/dL
  * Percent time below 54 mg/dL (superiority)

OTHER OUTCOMES:
CGM metrics related to hypoglycemia | 4-10 days
  - Percent <70 mg/dL
CGM metrics related to hypoglycemia | 4-10 days
  - Hypoglycemia events (defined as at least 15 consecutive minutes <54 mg/dL)
CGM metrics related to hyperglycemia | 4-10 days
  - Percent >300 mg/dL
CGM metrics related to hyperglycemia | 4-10 days
  - CGM-measured hyperglycemic events (≥90 minutes with glucose concentration >300 mg/dL in a 120min interval)
Glucose Variability | 4-10 days
  * glucose variability measured with the coefficient of variation
  * glucose variability measured with the standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Irl Hirsch, MD, Study Chair — University of Washington; Judy Sibayan, MPH, CCRP, Principal Investigator — Jaeb Center for Health Research; Roy Beck, MD, PhD, Study Director — Jaeb Center for Health Research
Locations (6):
- United States (6):
  - University of Colorado, Anschutz Inpatient Pavilion 1 and 2, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Baltimore Research and Education Foundation, Baltimore, Maryland
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Public data set will include the de-identified participants demographic and CGM data.
Supporting Information: Study Protocol
Time Frame: 1 year post completion
Access Criteria: Requests are entered on Jaeb Center for Health Research public website which collects name and contact information for individual requesting data along with reason for request, including planned analyses.
URL: http://public.jaeb.org

REFERENCES:
- [Background] Price CL, Hassi HO, English NR, Blakemore AI, Stagg AJ, Knight SC. Methylglyoxal modulates immune responses: relevance to diabetes. J Cell Mol Med. 2010 Jun;14(6B):1806-15. doi: 10.1111/j.1582-4934.2009.00803.x. Epub 2009 Jun 16. PMID 19538479
- [Background] Carey IM, Critchley JA, DeWilde S, Harris T, Hosking FJ, Cook DG. Risk of Infection in Type 1 and Type 2 Diabetes Compared With the General Population: A Matched Cohort Study. Diabetes Care. 2018 Mar;41(3):513-521. doi: 10.2337/dc17-2131. Epub 2018 Jan 12. PMID 29330152
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] NICE-SUGAR Study Investigators; Finfer S, Chittock DR, Su SY, Blair D, Foster D, Dhingra V, Bellomo R, Cook D, Dodek P, Henderson WR, Hebert PC, Heritier S, Heyland DK, McArthur C, McDonald E, Mitchell I, Myburgh JA, Norton R, Potter J, Robinson BG, Ronco JJ. Intensive versus conventional glucose control in critically ill patients. N Engl J Med. 2009 Mar 26;360(13):1283-97. doi: 10.1056/NEJMoa0810625. Epub 2009 Mar 24. PMID 19318384
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Van den Berghe G, Wilmer A, Hermans G, Meersseman W, Wouters PJ, Milants I, Van Wijngaerden E, Bobbaers H, Bouillon R. Intensive insulin therapy in the medical ICU. N Engl J Med. 2006 Feb 2;354(5):449-61. doi: 10.1056/NEJMoa052521. PMID 16452557
- [Background] Brunkhorst FM, Engel C, Bloos F, Meier-Hellmann A, Ragaller M, Weiler N, Moerer O, Gruendling M, Oppert M, Grond S, Olthoff D, Jaschinski U, John S, Rossaint R, Welte T, Schaefer M, Kern P, Kuhnt E, Kiehntopf M, Hartog C, Natanson C, Loeffler M, Reinhart K; German Competence Network Sepsis (SepNet). Intensive insulin therapy and pentastarch resuscitation in severe sepsis. N Engl J Med. 2008 Jan 10;358(2):125-39. doi: 10.1056/NEJMoa070716. PMID 18184958
- [Background] Preiser JC, Devos P, Ruiz-Santana S, Melot C, Annane D, Groeneveld J, Iapichino G, Leverve X, Nitenberg G, Singer P, Wernerman J, Joannidis M, Stecher A, Chiolero R. A prospective randomised multi-centre controlled trial on tight glucose control by intensive insulin therapy in adult intensive care units: the Glucontrol study. Intensive Care Med. 2009 Oct;35(10):1738-48. doi: 10.1007/s00134-009-1585-2. Epub 2009 Jul 28. PMID 19636533
- [Background] Davis GM, Spanakis EK, Migdal AL, Singh LG, Albury B, Urrutia MA, Zamudio-Coronado KW, Scott WH, Doerfler R, Lizama S, Satyarengga M, Munir K, Galindo RJ, Vellanki P, Cardona S, Pasquel FJ, Peng L, Umpierrez GE. Accuracy of Dexcom G6 Continuous Glucose Monitoring in Non-Critically Ill Hospitalized Patients With Diabetes. Diabetes Care. 2021 Jul;44(7):1641-1646. doi: 10.2337/dc20-2856. Epub 2021 Jun 7. PMID 34099515
- [Background] Galindo RJ, Migdal AL, Davis GM, Urrutia MA, Albury B, Zambrano C, Vellanki P, Pasquel FJ, Fayfman M, Peng L, Umpierrez GE. Comparison of the FreeStyle Libre Pro Flash Continuous Glucose Monitoring (CGM) System and Point-of-Care Capillary Glucose Testing in Hospitalized Patients With Type 2 Diabetes Treated With Basal-Bolus Insulin Regimen. Diabetes Care. 2020 Nov;43(11):2730-2735. doi: 10.2337/dc19-2073. Epub 2020 Jul 8. PMID 32641372
- [Background] Singh LG, Satyarengga M, Marcano I, Scott WH, Pinault LF, Feng Z, Sorkin JD, Umpierrez GE, Spanakis EK. Reducing Inpatient Hypoglycemia in the General Wards Using Real-time Continuous Glucose Monitoring: The Glucose Telemetry System, a Randomized Clinical Trial. Diabetes Care. 2020 Nov;43(11):2736-2743. doi: 10.2337/dc20-0840. Epub 2020 Aug 5. PMID 32759361
- [Background] Agarwal S, Mathew J, Davis GM, Shephardson A, Levine A, Louard R, Urrutia A, Perez-Guzman C, Umpierrez GE, Peng L, Pasquel FJ. Continuous Glucose Monitoring in the Intensive Care Unit During the COVID-19 Pandemic. Diabetes Care. 2021 Mar;44(3):847-849. doi: 10.2337/dc20-2219. Epub 2020 Dec 23. PMID 33361145
- [Background] Sadhu AR, Serrano IA, Xu J, Nisar T, Lucier J, Pandya AR, Patham B. Continuous Glucose Monitoring in Critically Ill Patients With COVID-19: Results of an Emergent Pilot Study. J Diabetes Sci Technol. 2020 Nov;14(6):1065-1073. doi: 10.1177/1932296820964264. Epub 2020 Oct 16. PMID 33063556
- [Background] Galindo RJ, Umpierrez GE, Rushakoff RJ, Basu A, Lohnes S, Nichols JH, Spanakis EK, Espinoza J, Palermo NE, Awadjie DG, Bak L, Buckingham B, Cook CB, Freckmann G, Heinemann L, Hovorka R, Mathioudakis N, Newman T, O'Neal DN, Rickert M, Sacks DB, Seley JJ, Wallia A, Shang T, Zhang JY, Han J, Klonoff DC. Continuous Glucose Monitors and Automated Insulin Dosing Systems in the Hospital Consensus Guideline. J Diabetes Sci Technol. 2020 Nov;14(6):1035-1064. doi: 10.1177/1932296820954163. Epub 2020 Sep 28. PMID 32985262
- [Background] Thomas C, Welsh JB, Lu S, Gray JM. Safety and Functional Integrity of Continuous Glucose Monitoring Components After Simulated Radiologic Procedures. J Diabetes Sci Technol. 2021 Jul;15(4):781-785. doi: 10.1177/1932296820920948. Epub 2020 Apr 22. PMID 32319318
- [Background] Critchley JA, Carey IM, Harris T, DeWilde S, Hosking FJ, Cook DG. Glycemic Control and Risk of Infections Among People With Type 1 or Type 2 Diabetes in a Large Primary Care Cohort Study. Diabetes Care. 2018 Oct;41(10):2127-2135. doi: 10.2337/dc18-0287. Epub 2018 Aug 13. PMID 30104296